CLINICAL TRIAL: NCT07083531
Title: Bone Loss, Physical Function and Frailty in Older Women With Sickle Cell Trait
Brief Title: Bone Loss, Physical Function and Frailty in Older Women With Sickle Cell Trait Sickle Cell Trait
Status: Recruiting | Type: Observational
Sponsor: UConn Health (Other)
Responsible Party: Principal Investigator, Biree Andemariam, Professor of Medicine, UConn Health
Other Study IDs: 22-327-1
Record Dates: First submitted 2024-06-24; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-03

CONDITIONS: Sickle Cell Disease; Sickle Cell Trait
Keywords: Sickle Cell Disease (SCD); Sickle Cell Trait (SCT)
MeSH Terms: conditions — Anemia, Sickle Cell; Sickle Cell Trait

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Once informed consent and HIPAA authorization are obtained, a certified member of the research staff will perform the venipuncture for CBC, hemoglobin electrophoresis, blood serum bone turnover markers, phosphate, calcium, and vitamin D analysis. Research participants will donate approximately 12-15 cc of whole blood via venipuncture.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Healthy volunteers without SCT: Healthy women of African descent at least 50 years old without sickle cell trait and who have not had a menstrual period for at least 12 consecutive months.
  Interventions: Other: Healthy volunteers without SCT
- Healthy volunteers with SCT: Healthy women of African descent at least 50 years old with sickle cell trait and who have not had a menstrual period for at least 12 consecutive months.
  Interventions: Other: Healthy volunteers with SCT

INTERVENTIONS:
Other: Healthy volunteers without SCT — Participants will donate blood for serum bone turnover markers, complete blood count, calcium, phosphorus, albumin, parathyroid hormone, and hemoglobin electrophoresis. Participants will undergo a bone density evaluation and muscle mass measurement via dual-energy x-ray absorptiometry (DEXA) scanning. Participants will fill out dietary calcium intake and pain burden questionnaires. Participants will fill out a survey for frailty assessment, undergo 6-minute walk gait velocity and short physical performance battery (SPPB).
  Groups: Healthy volunteers without SCT
Other: Healthy volunteers with SCT — Participants will donate blood for serum bone turnover markers, complete blood count, calcium, phosphorus, albumin, parathyroid hormone, and hemoglobin electrophoresis. Participants will undergo a bone density evaluation and muscle mass measurement via dual-energy x-ray absorptiometry (DEXA) scanning. Participants will fill out dietary calcium intake and pain burden questionnaires. Participants will fill out a survey for frailty assessment, undergo 6-minute walk gait velocity and short physical performance battery (SPPB).
  Groups: Healthy volunteers with SCT

SUMMARY:
This is a cross-sectional, clinical research study comparing postmenopausal women of African Descent (AD) with different hemoglobin genotypes: normal and sickle cell trait (SCT). This research study has two purposes. The first purpose is to determine whether having SCT is a risk factor for the development of bone thinning in older women. The second purpose is to investigate whether women with SCT have reduced muscle function and increased frailty compared to women without SCT. The investigators estimate enrolling 50 female volunteers who are at least 50 years old and have not had a menstrual period for at least 12 consecutive months. Volunteers need not know whether they have SCT as this will be evaluated as part of the study.

DETAILED DESCRIPTION:
This is a collaborative project involving three different disciplinary areas, including The Division of Hematology/Oncology, The Division of Endocrinology, and The Center on Aging (CoA)/Geriatrics in the UConn School of Medicine. The project consists of two specific aims: (1) determine effects of SCT on bone mineral density in postmenopausal women of African descent and (2) investigate the association of SCT on skeletal muscle function and frailty in postmenopausal women of African descent. The investigators hypothesize that individuals with SCT have reduced bone mineral density, decreased muscle function, and increased frailty compared to controls. This research may identify a hitherto unrecognized risk factor for racially disparate fracture incidence and outcomes in AD women. These findings will set the basis for a more extensive clinical study directly examining the association of SCT on fracture incidence and fracture-related morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Female of African Decent.
* Age 50 years or older.
* Lack of menstrual period for at least 12 consecutive months

Exclusion Criteria:

* Taking medications known to influence bone metabolism (e.g., glucocorticoids, hormonal therapy, cancer or chemotherapy meds, anti-resorptive medications or anabolic therapies).
* Known metabolic bone disorder (e.g., uncontrolled thyroid disease, hyperparathyroidism, Vitamin D deficiency)
* Taking an investigational drug
* Documented sickle cell disease

Min Age: 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Postmenopausal female volunteers of African Descent
Study Population: The target population includes healthy age-matched postmenopausal female volunteers of African Descent with and without SCT. Subjects will be eligible if they are at least 50 years old and have not had a menstrual period for at least 12 consecutive months.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-08-23 (Actual); Primary Completion 2025-08-23 (Estimated); Study Completion 2025-08-23 (Estimated)

PRIMARY OUTCOMES:
Difference in bone mineral density between older African descent (AD) women with (N=25) and without (N=25) sickle cell trait (SCT) | Day 1
  Particpants will undergo dual energy xray absorptiometry.

SECONDARY OUTCOMES:
Difference in 25-OH vitamin D between older African descent (AD) women with (N=25) and without (N=25) sickle cell trait (SCT) | Day 1
  Participants will undergo blood testing to measure 25-OH Vitamin D levels in nanograms per milliliter.
Difference in calcium between older African descent (AD) women with (N=25) and without (N=25) sickle cell trait (SCT) | Day 1
  Participants will undergo blood testing to measure calcium levels in milligrams per deciliter.
Difference in parathyroid hormone between older African descent (AD) women with (N=25) and without (N=25) sickle cell trait (SCT) | Day 1
  Participants will undergo blood testing to measure parathyroid hormone levels in picograms per milliliter.
Effect of sickle cell trait (SCT) on frailty in older African descent (AD) women | Day 1
  Participants will have frailty assessed using both the Fried phenotype and the Rockwood Frailty Index.
Effect of sickle cell trait (SCT) on muscle mass in older African descent (AD) women | Day 1
  Particpants will undergo dual energy xray absorptiometry to assess muscle mass.
Effect of sickle cell trait (SCT) on muscle function in older African descent (AD) women. | Day 1
  Participants will undergo a 6-minute walk and gait velocity. In addition, the short physical performance battery (SPPB) will be measured. The SPPB is an objective assessment tool for evaluating lower extremity functioning in older persons, balance, lower extremity strength, and functional capacity.

CONTACTS AND LOCATIONS:
Overall Officials: Biree Andemariam, MD, Principal Investigator — UConn Health
Locations (1):
- UConn Health, Farmington, Connecticut, United States